CLINICAL TRIAL: NCT06843096
Title: Contrast-Enhanced Mammography (CEM) in the Evaluation of Cancer of Unknown Primary Syndrome (CUP): A Multicentric Observational Study
Brief Title: Contrast Enhanced Mammography in the Evaluation of Cancer of Unknown Primary Syndrome
Acronym: CEM_CUP_syndr
Status: Enrolling by invitation | Type: Observational
Sponsor: Graziella di Grezia (Other)
Collaborators: Link Campus University (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor-Investigator, Graziella di Grezia, Principal Investigator, Link Campus University
Organization: Link Campus University (Other)
Other Study IDs: T_1_2025
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Diagnosis; Breast Cancer Prevention
Keywords: Contrast-Enhanced Mammography (CEM); Cancer of Unknown Primary (CUP); Breast Cancer; MRI (Magnetic Resonance Imaging); Diagnostic Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Mammography (CEM) — The intervention in this study involves Contrast-Enhanced Mammography (CEM), a specialized imaging technique that combines standard mammography with contrast-enhanced imaging to detect neo-angiogenesis, which is a characteristic of malignancy. Unlike traditional mammography, CEM utilizes both low-energy and high-energy images to provide enhanced visualization of tissue vascularity, aiding in the identification of occult primary tumors, particularly in patients with Cancer of Unknown Primary (CUP) syndrome.
  Patients who present with CUP syndrome, suspected of having a primary breast malignancy, will undergo CEM as part of their diagnostic workup. The CEM findings will be compared with other conventional imaging modalities, including ultrasound and MRI, to assess the diagnostic accuracy of CEM in detecting primary breast tumors. The intervention will also involve correlating the imaging results with histopathological findings from biopsy or surgical specimens.
  This study aims to demons

SUMMARY:
This study aims to evaluate the role of Contrast-Enhanced Mammography (CEM) in identifying the primary tumor site in patients presenting with Cancer of Unknown Primary (CUP) syndrome. By integrating functional and anatomical imaging, the study explores CEM's diagnostic value compared to standard imaging modalities in a single-center setting.

DETAILED DESCRIPTION:
The study of CUP syndrome was conducted with MRI, but we propose the study with CEM

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients aged 18 years or older.
* Diagnosis of CUP: Patients with a clinical diagnosis of Cancer of Unknown Primary (CUP) syndrome.
* Suspected Breast Malignancy: Patients with clinical or imaging suspicion of a primary breast malignancy.
* Informed Consent: Patients who are able to provide informed consent to participate in the study.
* Presence of Breast Tissue: Female or transgender patients with breast tissue eligible for Contrast-Enhanced Mammography (CEM).

Exclusion Criteria:

* Confirmed Primary Tumor: Patients with a confirmed primary tumor identified in an organ other than the breast.
* Contraindications to Contrast Agents: Patients with contraindications to the use of iodinated contrast agents (e.g., severe allergic reactions to contrast).
* Severe Renal Impairment: Patients with severe renal impairment (eGFR < 30 mL/min/1.73 m²) who cannot safely receive contrast agents.
* Pregnancy or Breastfeeding: Pregnant or breastfeeding women, as contrast administration may be harmful to the fetus or neonate.
* Severe Medical Conditions: Patients with severe medical conditions that may compromise their participation or safety in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to cisgender women and transgender women who have breast tissue and are presenting with Cancer of Unknown Primary (CUP) syndrome and suspected primary breast malignancy. Individuals must have mammary tissue to be eligible for participation, as the study involves Contrast-Enhanced Mammography (CEM), which is specifically used to evaluate breast malignancies.
Study Population: The study population will consist of adult patients (aged 18 years and older) who are diagnosed with Cancer of Unknown Primary (CUP) syndrome and are suspected of having a primary breast malignancy based on clinical presentation or imaging findings. Eligible patients will have breast tissue suitable for Contrast-Enhanced Mammography (CEM) and will undergo CEM as part of their diagnostic workup to evaluate the potential primary tumor site.
  The population will be diverse in terms of age, race, and ethnic backgrounds, provided they meet the inclusion criteria and do not fall under any of the exclusion criteria listed.
  The study aims to include a cohort of patients with different stages of CUP syndrome to evaluate the effectiveness of CEM in identifying hidden primary tumors and its impact on clinical management and treatment decisions.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of Primary Tumors using Contrast-Enhanced Mammography (CEM) in Patients with CUP Syndrome | From enrollment to the end of treatment at 12 months
  The primary outcome of this study is the detection rate of primary tumors in patients presenting with Cancer of Unknown Primary (CUP) syndrome using Contrast-Enhanced Mammography (CEM). The detection rate will be determined by comparing the CEM findings with histopathological results from biopsies or surgical specimens. This will allow us to assess the diagnostic accuracy of CEM in identifying occult primary tumors, particularly in the context of breast cancer.

SECONDARY OUTCOMES:
Sensitivity, Specificity, and Diagnostic Accuracy of CEM compared to Standard Imaging Modalities (Ultrasound, MRI, Mammography) | From enrollment to the end of treatment at 12 months
  This secondary outcome aims to evaluate the sensitivity, specificity, and diagnostic accuracy of CEM in detecting primary tumors compared to other conventional imaging techniques, including ultrasound, MRI, and standard mammography. These metrics will be analyzed to determine the relative effectiveness of CEM as a diagnostic tool.
Correlation of CEM Findings with Histopathological Results | From enrollment to the end of treatment at 12 months
  This measure aims to correlate the CEM findings with the histopathological results from biopsy or surgical specimens. This will assess how well the CEM images match the final diagnosis of primary tumors based on tissue analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Di Grezia, medicine and surgery, Principal Investigator — Link Campus University
Locations (1):
- Link Campus University, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided